CLINICAL TRIAL: NCT00020358
Title: Randomized Comparison of Three Schedules of Peptide Immunization in Patients With Stage II or III, or Completely Resected Metastatic Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068299; NCI-00-C-0216; NCI-2391; NCT00006287 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2003-03

CONDITIONS: Melanoma (Skin)
Keywords: stage I melanoma; stage II melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; incomplete Freund's adjuvant

INTERVENTIONS:
Biological: aldesleukin
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: tyrosinase peptide

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Vaccine therapy may be an effective treatment for melanoma.

PURPOSE: Randomized phase II trial to study the effectiveness of three vaccine therapy regimens in treating patients who have melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the immunologic activity of three different schedules of peptide immunization with gp100:209-217 (210M) or gp100:17-25 antigen and tyrosinase:368-376 (370D), tyrosinase:240-251 (244S), tyrosinase:206-214 (closed to accrual 11/05/01), or tyrosinase-related protein-1 (ORF3):1-9 peptide (closed to accrual 11/05/01) emulsified in Montanide ISA-51 in patients with melanoma at high risk for recurrence.
* Compare the response rate to treatment with interleukin-2 (IL-2) after being immunized with this regimen with the usual response rate to IL-2 in this patient population.
* Determine whether an exploratory cohort of HLA-A2-positive patients demonstrate immunologic activity to immunization with 2 peptides emulsified together.

OUTLINE: This is a randomized study. Patients are stratified according to HLA type (A0201 vs A1 vs A3 vs A24 vs A31). (HLA-A24 and HLA-A31 closed to accrual 11/05/01). Patients are randomized to 1 of 3 treatment arms and are given an assigned vaccine, which is emulsified in Montanide ISA-51.

* HLA typing:

  * HLA-A2: gp100:209-217 (210M) and tyrosinase:368-376 (370D)
  * HLA-A1: tyrosinase:240-251 (244S)
  * HLA-A3: gp100:17-25
  * HLA-A24: tyrosinase:206-214 (closed to accrual 11/05/01)
  * HLA-A31: tyrosinase-related protein-1 (ORF3):1-9 (closed to accrual 11/05/01)
* Arm I: Patients receive assigned vaccine subcutaneously (SC) weekly for 10 weeks followed by 3 weeks of no treatment.
* Arm II: Patients receive assigned vaccine SC on days 1, 22, 43, and 64.
* Arm III: Patients receive assigned vaccine SC on days 1-4, 22-25, 43-46, and 64-67.

Treatment in all arms repeats every 13 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

After the completion of the randomized arms of HLA-A2 patients, additional HLA-A2 patients receive immunization with gp100:209-217 (210M) and tyrosinase:368-376 (370D) emulsified in Montanide ISA-51 SC once every 3 weeks for 4 courses.

Patients with progressive disease may receive interleukin-2 IV over 15 minutes every 8 hours for up to 4 days. Treatment repeats every 10-14 days for at least 4 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease or mixed or partial response to treatment may receive additional courses every 2 months.

Patients are followed at 6 months.

PROJECTED ACCRUAL: A total of 324 patients (19-33 per arm for the HLA-A0201 stratum, 13-16 per arm for the other 4 strata, and 33 per the additional HLA-A2 cohort) will be accrued for this study within 2 years. (HLA-A24 and HLA-A31 closed to accrual 11/05/01).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of melanoma, including one of the following characteristics:

  * Lesions at least 1.5 mm in thickness
  * At least 1 positive lymph node
  * Ulcerated lesion
  * Local recurrence
  * Metastatic lesions completely resected within the past 6 months
* Clinically disease free within the past 6 weeks
* HLA-A1, A3, A24, A31, or 0201 positive (HLA-A24 and HLA-A31 closed to accrual 11/05/01)
* No ocular or mucosal melanoma

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 90,000/mm^3

Hepatic:

* Bilirubin no greater than 1.6 mg/dL (3.0 mg/dL in Gilbert's syndrome)
* AST and ALT less than 3 times normal
* Hepatitis B surface antigen negative

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* For interleukin-2 (IL-2) therapy:

  * No cardiac ischemia, myocardial infarction, or cardiac arrhythmias
  * Stress cardiac test required if abnormal EKG, symptoms of cardiac ischemia or arrhythmia, or older than 50 years

Pulmonary:

* For IL-2 therapy:

  * No obstructive or restrictive pulmonary disease
  * FEV_1 greater than 60% predicted if prolonged history of cigarette smoking or symptoms of respiratory dysfunction

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No active systemic infections, autoimmune disease, or active primary or secondary immunodeficiency

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior systemic biologic therapy for melanoma
* No prior gp100 antigen or tyrosinase or TRP-1 peptide
* No other concurrent systemic biologic therapy for melanoma

Chemotherapy:

* At least 3 weeks since prior systemic chemotherapy and recovered
* No concurrent systemic chemotherapy for melanoma

Endocrine therapy:

* At least 3 weeks since prior systemic endocrine therapy for melanoma
* No concurrent systemic steroid therapy

Radiotherapy:

* At least 3 weeks since prior systemic radiotherapy and recovered
* No concurrent systemic radiotherapy for melanoma

Surgery:

* See Disease Characteristics

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-09; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Rosenberg SA, Sherry RM, Morton KE, Scharfman WJ, Yang JC, Topalian SL, Royal RE, Kammula U, Restifo NP, Hughes MS, Schwartzentruber D, Berman DM, Schwarz SL, Ngo LT, Mavroukakis SA, White DE, Steinberg SM. Tumor progression can occur despite the induction of very high levels of self/tumor antigen-specific CD8+ T cells in patients with melanoma. J Immunol. 2005 Nov 1;175(9):6169-76. doi: 10.4049/jimmunol.175.9.6169. PMID 16237114